CLINICAL TRIAL: NCT04886778
Title: Efficacy and Safety of Low-Carbohydrate Diet Combined With Probiotics for Weight Loss in Male Obese Patients.：A Randomized, Double-blind, Placebo, Controlled Clinical Trial.
Brief Title: Efficacy and Safety of Low-Carbohydrate Diet Combined With Probiotics for Weight Loss in Male Obese Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Jia (Other)
Responsible Party: Sponsor-Investigator, Sun Jia, Vice-Chairman of the Department of Endocrinology and Metabolism，Chief Physician，Associate Professor，Doctor Supervisor of Endocrinology, Zhujiang Hospital
Organization: Zhujiang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021LX0021_GY
Record Dates: First submitted 2021-05-01; First posted 2021-05-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Obesity
Keywords: Carbohydrate-restricted diet; Probiotics; Efficacy and safety; Low-carbohydrate diet; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: 44 obese participants who meet the inclusion/exclusion criteria are randomly assigned to group A and group B at a ratio of 1:1. As the experimental group, group A was treated with a 12-week low-carbohydrate diet combined with probiotic compound preparations, and group B was treated as a control group with a 12-week low-carbohydrate diet combined with placebo treatment. Since the probiotic compound preparation is made of Lactobacillus reuteri, Lactobacillus gasseri, Lactobacillus acidophilus, Bifidobacterium lactis and resistant dextrin (water soluble dietary fiber), in order to eliminate the effect of resistant dextrin (water-soluble meal fiber) on the experimental results, the placebo is prepared from resistant dextrin (water-soluble meal fiber) and is packaged to be consistent with the appearance of the probiotic compound preparation.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A or Trial group (Experimental): Group A was treated with a 12-week low-carbohydrate diet combined with probiotic compound preparations.
  Interventions: Dietary Supplement: Low-carbohydrate diet; Dietary Supplement: Probiotic compound preparations
- Group B or Placebo control group (Placebo Comparator): Group B was treated as a control group with a 12-week low-carbohydrate diet combined with placebo treatment.
  Interventions: Dietary Supplement: Low-carbohydrate diet; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Low-carbohydrate diet — Participants will be instructed to maintain a daily dietary energy intake of less than 1600 kcal.Based on the low-carbohydrate diet model, the proportion of daily intake of carbohydrate was about 30%, and this ratio was up to 30%, 40% of protein and fat respectively.Participants should choose unprocessed whole grains, potatoes, vegetables, meat, fish, eggs, soy products, sugar-free dairy products, designated varieties of low-GI fruits and nuts, etc. as breakfast, and avoid processed meats and high-fat red meat and poultry skins. Standard nutritious meal instead of daily lunch and dinner meals, that is to say, participants should take one nutritional bar for lunch and dinner (310 kcal totally, provided by Guangzhou Nanda Fett Nutrition and Health Consulting Co., Ltd.), and avoid starchy foods. Other food varieties are required to be the same as breakfast. Plant oil is the main cooking oil, and participants will be instructed to drink 2L water every day.
Dietary Supplement: Probiotic compound preparations — The probiotic compound preparation，named Junyi Yili® Probiotics，is made of Lactobacillus reuteri, Lactobacillus gasseri, Lactobacillus acidophilus and Bifidobacterium lactis, and resistant dextrin contained water-soluble dietary fiber. The subjects will take this probiotic compound preparations with purified water after three meals every day, 1 sachet each time.
  Other Names: Junyi Yili® Probiotics
  Arms: Group A or Trial group
Dietary Supplement: Placebo — Placebo is made of resistant dextrin which contained water-soluble dietary fiber. The subjects were taken this placebo with purified water after three meals every day, 1 sachet each time.
  Arms: Group B or Placebo control group

SUMMARY:
Over the years, increasing obesity prevalence represents an important threat to national and global public health. Many strategies studied for weight loss have reported that low-carbohydrate diets showed beneficial effects on weight loss for obese patients. However, individual weight losses have varied widely within low-carbohydrate diet groups due to the influence of gut microbiota, which was found in the previous clinical studies of our team (ChiCTR1800015156). Numerous animal studies and clinical trials have evaluated the impact of probiotics on glucose and lipid metabolism as well as weight-loss interventions. However, the effect of the different probiotic strains may play a different role in the same species. Therefore, our team isolated new strains (Lactobacillus reuteri PLBK1，GDMCC No: 60828、Lactobacillus reuteri PLBK2，GDMCC No: 60829、Lactobacillus gasseri PLBK3，GDMCC No: 60830、Lactobacillus acidophilus PLBK4，GDMCC No: 60831、Bifidobacterium lactis PLBK5，GDMCC No: 60832) from the oral cavity, feces or environment of the Chinese race in the previous study. The mixed solid beverage composed of these five strains has local characteristics and meets the requirements of the national standard for food additives, which has obtained the national food production license (SC10632028100205).In our previous animal experiments, the treatment of compound preparation of the above five strains improve insulin resistance and dyslipidemia effectively in obese mice induced by high-fat diet，which obtained significant weight loss . Nevertheless, clinical trials are needed to be carried out to confirm its clinical effect. Therefore, we aimed to conduct a randomized, double-blind, placebo-controlled prospective study on the basis of previous research. In order to evaluate the efficacy and safety, as well as the effect on glucose and lipid metabolism of low-carbohydrate diet combined with probiotics in obese participants, the study will last for 12 weeks. At the same time, Magnetic Resonance Imaging (MRI) will be used to clarify change in body fat distribution, which may provide more clinical evidence for the application of this program in the prevention and treatment of obesity in the future.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial. According to the preliminary experimental results, the decrease in weight of the experimental group intervening by low-carbohydrate diet combined with probiotics compound preparation was up to (6.5±1.1) kg over the whole study period compared to that in control group adopted low-carbohydrate diet combined with placebo, which was about (4.1±0.8) kg. When taking superiority cutoff (δ) of 1.5kg, in α = 0.025 (one-sided) and the power (1-β) = 0.8, on the premise that the two groups of research objects are equal in number, the sample size of the experimental group and the control group is 19 cases respectively by using the PASS11.0 software to calculate (N1=N2=19 cases). Considering that a dropout rate of no more than 10% may occur during follow-up, this study included a total sample size of no less than 44.

Forty-four obese participants who meet the inclusion/exclusion criteria are randomly assigned to group A and group B at a ratio of 1:1. As the trial group, group A was treated with a 12-week low-carbohydrate diet combined with probiotic compound preparations, and group B was treated as a placebo control group with a 12-week low-carbohydrate diet combined with placebo treatment. Since the probiotic compound preparation is made of Lactobacillus reuteri, Lactobacillus gasseri, Lactobacillus acidophilus, Bifidobacterium lactis, and resistant dextrin (water-soluble dietary fiber), to eliminate the effect of resistant dextrin (water-soluble meal fiber) on the experimental results, the placebo is prepared from resistant dextrin (water-soluble meal fiber) and is packaged to be consistent with the appearance of the probiotic compound preparation.

During the trial period, participants will attend face-to-face visits at 4-week (visit 3), 8-week (visit 4), and 12-week (visit 5). During each follow-up visit, participants will be asked about their dietary structure, average daily calorie intake, exercise volume, adverse events, and so on. Research assistants will record their heart rate, blood pressure, height, weight, BMI, waist circumference, and waist-to-hip ratio. During the 12-week (visit 5), research assistants will record fasting blood glucose, fasting insulin, insulin resistance index (HOMA-IR), biomarkers of lipids metabolism (TG/TC/LDL/HDL), subcutaneous fat and visceral fat volume, the fat fraction (FF). Fecal samples will be collected by participants at baseline as well as at the end stage and be divided into 10 parts, each one is about 200-300mg. All fecal samples will be stored in a -80 ℃ freezer by researchers. At the end of the experiment, fecal samples will be uniformly sent to Metabo-Profile Biotechnology (Shanghai) Co., Ltd. to detect the composition of gut microbes.

The data of this project will be collected from the Department of Endocrinology and Metabolism, Zhujiang Hospital of Southern Medical University. Relevant information will be obtained by consulting the inspection system and asking patients. All data will be recorded independently by two specialized statisticians.

Data management strictly abides by relevant regulations, and any transfer of electronic data or subject-related data must be approved by the data management department. In case data is transmitted through non-secure electronic networks, corresponding data protection rules must be followed.

The statistical methods are as follow:

1. General analysis: In this study, if no special instructions are given, the data will be described and analyzed according to the following general principles. Statistics description: The mean, standard deviation and confidence interval will be given in measurement data, and if necessary, the minimum, maximum, P25, median and P75 will be given. When the non-parametric method is used, the median and interquartile range will be given. The frequency distribution and the corresponding percentage will be given in counting data. The frequency distribution and the corresponding percentage and average rank will be given in grade data. Basic principles: All statistical inferences use two-sided tests, the statistically significant test level is set at 0.05, and the confidence interval of the parameters is estimated to be 95% confidence interval. The comparison of counting data between groups depends on the theoretical frequency, using χ2 test, continuous correction χ2 test or Fisher's exact probability method. Two independent sample T-tests is used to compare normally distributed baseline measurement data between groups. For non-normal distribution baseline measurement data, the Wilcoxon rank sum test is used for comparison between groups. Continuous variables measured at multiple time points are analyzed using a Mixed effect model. p<0.05 is considered significant in the study. Missing data: The mixed linear model will be used to obtain the point estimation and standard deviation of the treatment effect. The Markov chain Monte Carlo method is used to fill in the missing data in the multivariate analysis. Abnormal data: Interquartile range whose observation value is greater than P75 or less than P25 more than 3 times will be judged as outlier data. In the analysis process, sensitivity analysis will be used for outlier data, that is, both retention and elimination of outlier data are analyzed. If the results are not contradictory, the data will be retained; if contradictory, it will be depended on the specific situation.
2. Basic characteristics: The mean, standard deviation, median, maximum and minimum will be calculated for quantitative data such as age, height, weight and BMI. The frequency and percentage will be listed for qualitative information such as gender.
3. Efficacy analysis: The efficacy analysis will be based on the Full Analysis Set (FAS). Analysis of the main efficacy indicators: the extent of weight loss during the trial period is a continuous variable, so that the results will be analyzed using Mixed effects model. In the model, subject factors are considered as random effects and intervention, time and mutual interaction effects are considered as fixed effects.Analysis of secondary efficacy indicators: After 12-week intervention, the continuous variables such as insulin resistance indicators, waist circumference, waist-to-hip ratio, lipids (TG/TC/LDL/HDL), body fat percentage (BF%), subcutaneous and visceral adipose tissue volume, fat fraction (FF) compared with the baseline will be analyzed by mixed effects model. Other categorical variables are analyzed using χ2 test, continuous correction χ2 test or Fisher's exact probability method.
4. Security analysis: The safety rating will be based on the safety set (SS), with descriptive statistical analysis as the main focus. The adverse events, serious adverse events and reactions occurred in the two groups will be analyzed. An adverse reaction is defined as an adverse event that has a relationship with the study drug as "definitely related or may be related or undeterminable". The laboratory results that are normal before the trial but abnormal after treatment will be described. The mean, standard deviation, median, minimum and maximum values of blood pressure, heart rate and laboratory indicators before and after the intervention in the two groups, as well as the number and rate of "normal turned abnormal" or "abnormal aggravation" of vital signs and laboratory indicators will be calculated.
5. Sensitivity analysis: Sensitivity analysis will be performed after missing data filling and abnormal data elimination.
6. Statistical software and general requirements: SPSS 24.0 statistical software is used for data entry and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male;
* 18 to 35 years old;
* BMI≥28kg/m2;
* No contraindications for MRI examination;
* No alcohol intake, no use of any probiotic-related foods or medications, antibiotics, hormones and weight-loss products in the past three months;
* No other metabolic diseases;
* Volunteering to participate in and cooperate with the research and sign the written informed consent.

Exclusion Criteria:

* Subjects suffered from Secondary obesity including hypercortisolism, hypothyroidism, insulinoma, drug-induced obesity, etc.
* Obesity-related complications that may be life-threatening or cause serious consequences in the short term have occurred.
* Any of the following cardiovascular diseases have occurred in the past：

  1. Myocardial infarction.
  2. Cerebral infarction.
  3. Cardiac or revascularization surgery such as coronary artery bypass graft surgery and percutaneous transluminal coronary angioplasty.
  4. Unstable angina pectoris;
  5. Congestive heart failure diagnosed as Class III or IV of the New York Heart Association.
  6. Transient ischemic attack or significant cerebrovascular disease.
* Patients with symptoms of gastrointestinal diseases, including intestinal obstruction, intestinal ulcer and gastrointestinal bleeding.
* A history of gastrointestinal surgery, such as bariatric surgery, banding surgery, gastrointestinal anastomosis and enterectomy.
* A state of known immunodeficiency, including but not limited to individuals who have experienced organ transplantation or acquired immunodeficiency syndrome (AIDS).
* Subjects who cannot comply with the protocol and patients with serious physical or psychological diseases that may affect the effectiveness or safety under the judgment of the investigator.
* Patients who cannot cooperate to complete the entire intervention and follow-up due to various other factors.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in body weight. | At 12th week after the intervention.
  When measuring height, the subjects are required to take off their shoes, hats, and coats, keep their feet together in an upright position, keep their shoulders, head, and heels close to the ruler, and look straight ahead with the right-angle plate close to the top of the head. The measurement standard of height is accurate to 0.1cm. When measuring body weight, the subjects are required to take off their shoes, hats, and single clothes for measurement and the measurement standard of body weight is accurate to 0.1kg. Body mass index (BMI) is calculated by dividing body weight (kg) by the square of height (m2). All measurements will be performed by trained staff.
Incidence rate of adverse events. | Up to 12 weeks.
  During the trial period, participants will attend several times face-to-face visits. At other times, participants will be contacted by investigators by phone to supervise their diets, to ensure compliance, to record observed side effects and adverse events in time.

SECONDARY OUTCOMES:
Phased changes in body weight at 4th and 8th weeks. | At 4th and 8th weeks after the intervention.
  When measuring body weight, the subjects are required to take off their shoes, hats, and single clothes for measurement and the measurement standard of body weight is accurate to 0.1kg. All measurements are performed by trained staff.
Phased changes in body mass index at 4th and 8th weeks. | At 4th and 8th weeks after the intervention.
  When measuring height, the subjects are required to take off their shoes, hats, and coats, keep their feet together in an upright position, keep their shoulders, head, and heels close to the ruler, and look straight ahead with the right-angle plate close to the top of the head. The measurement standard of height is accurate to 0.1cm. When measuring body weight, the subjects are required to take off their shoes, hats, and single clothes for measurement and the measurement standard of body weight is accurate to 0.1kg. Body mass index (BMI) is calculated by dividing body weight (kg) by the square of height (m2). All measurements are performed by trained staff.
Changes in fasting blood glucose. | At 12th week after the intervention.
  Fasting blood glucose will be uniformly implemented in the Laboratory of Zhujiang Hospital.
Changes in fasting insulin. | At 12th week after the intervention.
  Fasting insulin will be uniformly implemented in the Laboratory of Zhujiang Hospital.
Changes in insulin resistance index (HOMA-IR) . | At 12th week after the intervention.
  The steady-state model assessment method will be used to calculate homeostasis model assessment of insulin resistance (HOMA-IR): HOMA-IR= fasting blood glucose (mmol/L) × fasting insulin (mIU/L)/22.5.
Changes in waist circumference. | At 4th, 8th and 12th week after the intervention.
  When measuring the waist circumference, the subjects were required to wear thin underwear, and the researchers used a soft ruler to measure the circumference of a circle around the umbilicus, and the measurement of waist circumference was accurate to 0.1cm. All measurements are performed by trained staff.
Changes in waist-to-hip ratio. | At 4th, 8th and 12th week after the intervention.
  When measuring the waist circumference, the subjects were required to wear thin underwear, and the researchers used a soft ruler to measure the circumference of a circle around the umbilicus, and the measurement of waist circumference was accurate to 0.1cm. When measuring the hip circumference, the subjects are required to wear thin underwear, and a soft ruler is required to measure the circumference of the most protruding part backwards around the buttocks to the nearest 0.1cm. The waist-to-hip ratio is calculated by dividing the waist circumference (cm) by the hip circumference. All measurements are performed by trained staff.
Changes in triglycerides in the blood. | At 12th week after the intervention.
  Blood triglycerides will be tested by the Laboratory of Zhujiang Hospital.
Changes in total cholesterol in the blood. | At 12th week after the intervention.
  Blood total cholesterol will be tested by the Laboratory of Zhujiang Hospital.
Changes in low-density lipoprotein in the blood. | At 12th week after the intervention.
  Blood low-density lipoprotein will be tested by the Laboratory of Zhujiang Hospital.
Changes in high-density lipoprotein in the blood. | At 12th week after the intervention.
  Blood high-density lipoprotein will be tested by the Laboratory of Zhujiang Hospital.
Changes in body fat percentage（BF%）. | At 12th week after the intervention.
  Body fat percentage will be tested using an IOI353 body composition analyzer manufactured by Jawon Medica in Korea. Before the measurement, the subjects will be required to have an empty stomach and instructed to empty their urine and bowels. The subjects will be asked to use 75% alcohol gauze to wipe their hands and feet to make them fully contact the electrode surface of the analyzer after taking off their socks. Then researchers having training before will enter the patient's personal information on the body composition analyzer computer, and press the finish and start buttons next to get the body fat percentage (BF%) measurement result.
Changes in subcutaneous fat volumn. | At 12th week after the intervention.
  After a period of adaptation, the subjects will be performed MRI scans on the their abdomen and pelvis in the MR room of Zhujiang Hospital of Southern Medical University at a fixed ambient temperature，operated by researchers using the 3.0T MRI scanner Ingenia which was made by Philips in (the) Netherlands to . The six-echo 3D gradient echo DIXON sequence (mDixon Quant, Philips Healthcare) will be used to scan. The water, fat, proton density fat fractions (PDFF) and T2*mapping images can be obtained through the algorithms. Based on the open-source image processing software "3D Slicer" of Harvard Medical School, the fat images is semiautomatically segmented and the segmentation range is defined from the lower edge of the T9 vertebral body to the upper edge of the bilateral femoral head. The subcutaneous adipose (SAT) volumn can be obtained respectively.
Changes in visceral adipose volume. | At 12th week after the intervention.
  After a period of adaptation, the subjects will be performed MRI scans on the their abdomen and pelvis in the MR room of Zhujiang Hospital of Southern Medical University at a fixed ambient temperature，operated by researchers using the 3.0T MRI scanner Ingenia which was made by Philips in (the) Netherlands to . The six-echo 3D gradient echo DIXON sequence (mDixon Quant, Philips Healthcare) will be used to scan. The water, fat, proton density fat fractions (PDFF) and T2*mapping images can be obtained through the algorithms. Based on the open-source image processing software "3D Slicer" of Harvard Medical School, the fat images is semiautomatically segmented and the segmentation range is defined from the lower edge of the T9 vertebral body to the upper edge of the bilateral femoral head. The visceral adipose volume can be obtained respectively.
Changes in fat fraction (FF). | At 12th week after the intervention.
  After a period of adaptation, the subjects will be performed MRI scans on the their abdomen and pelvis in the MR room of Zhujiang Hospital of Southern Medical University at a fixed ambient temperature，operated by researchers using the 3.0T MRI scanner Ingenia which was made by Philips in (the) Netherlands to . The six-echo 3D gradient echo DIXON sequence (mDixon Quant, Philips Healthcare) will be used to scan. The water, fat, proton density fat fractions (PDFF) and T2*mapping images can be obtained through the algorithms. Based on the American open-source image processing software "ITK-SNAP", an ROI with a diameter of about 20mm can be drawn on each hepatic segment on the PDFF images, and the average value will represent the liver fat fraction(FF).
Changes in gut microbe composition. | At 12th week after the intervention.
  At baseline as well as at the end of the trial, researcher will collect participants' fecal samples and divided into 10 portions that each one is about 200-300mg, all of which will be frozen and stored in the refrigerator at -80 ℃. At the end of the experiment, the fecal samples will be uniformly sent to Metabo-Profile Biotechnology (Shanghai) Co., Ltd. to detect the composition of gut microbes.
Changes in gut microbe relative abundance. | At 12th week after the intervention.
  At baseline as well as at the end of the trial, researcher will collect participants' fecal samples and divided into 10 portions that each one is about 200-300mg, all of which will be frozen and stored in the refrigerator at -80 ℃. At the end of the experiment, the fecal samples will be uniformly sent to Metabo-Profile Biotechnology (Shanghai) Co., Ltd. to detect the relative abundance of gut microbes.
Phased incidence rate of adverse event. | At 4th, 8th week after the intervention.
  The investigator will ask participants in face-to-face visits or contacted with them by phone to record observed side effects and adverse events in time.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Sun, MD,PhD, Study Chair — Zhujiang Hospital; Hong Chen, MD,PhD, Principal Investigator — Zhujiang Hospital; Zhen Zhang, MD,PhD, Principal Investigator — Zhujiang Hospital; Zhibo Wen, MD,PhD, Principal Investigator — Zhujiang Hospital; Yuting Ruan, MD,PhD, Principal Investigator — Zhujiang Hospital; Jitong Li, MD,PhD, Principal Investigator — Zhujiang Hospital; Qing Yang, MN, Principal Investigator — Zhujiang Hospital
Locations (1):
- The Pearl River Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No